CLINICAL TRIAL: NCT05668715
Title: Comparison of the Efficacy of Transcutaneous Tibial Nerve Stimulation in Antimuscarinic Naive and Refractory Women With Idiopathic Overactive Bladder
Brief Title: Transcutaneous Tibial Nerve Stimulation in Antimuscarinic Naive and Refractory Women With Idiopathic Overactive Bladder
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Pamukkale University (Other)
Responsible Party: Principal Investigator, Necmettin Yildiz, Professor Doctor, Pamukkale University
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: pamukkaleu.ftr.NYildiz.001
Record Dates: First submitted 2022-11-30; First posted 2022-12-30 (Actual); Last update posted 2022-12-30 (Actual); Status verified 2022-12

CONDITIONS: Urinary Bladder, Overactive
MeSH Terms: conditions — Urinary Bladder, Overactive

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1: Antimuscarinic Naive (AM-N) (Experimental): None of the women had previously taken anti-muscarinic agents and oral ß3 adrenoreceptor agonist (mirabegron) in this group.
  Interventions: Other: Transcutaneous tibial nerve stimulation (TTNS)
- Group 2: Antimuscarinic Refractory (AM-R) (Active Comparator): Women with idiopathic OAB refractory to anti-muscarinic agents and oral ß3 adrenoreceptor agonist (mirabegron) when 2 or more were administered for at least 6 weeks each and failure was due to lack of efficacy with or without side effects were included in this group.
  Interventions: Other: Transcutaneous tibial nerve stimulation (TTNS)

INTERVENTIONS:
Other: Transcutaneous tibial nerve stimulation (TTNS) — PTNS has some disadvantages such as it is a minimally invasive method applied by needle, and the need to go to the hospital for this. However, the number of studies on transcutaneous tibial nerve stimulation (TTNS) (non-invasive and can be applied at home) tends to increase in recent years

SUMMARY:
In this study is the first prospective trial that compares the efficacy of TTNS in antimuscarinic naive and refractory women with idiopathic OAB. In this study, it was aimed to compare the effectiveness of TTNS on quality of life (QoL) and clinical parameters related to OAB in antimuscarinic naive and refractory women. The results of this study would make it easier to understand the place of TTNS among the treatment options in women with idiopathic OAB.

DETAILED DESCRIPTION:
This study was planned as a prospective clinical trial. The trial was carried out in the Urogynecological Rehabilitation Unit of Physical Medicine and Rehabilitation Department, in between January 2023 and June 2023. The local ethics committee approved the study. All women were informed about the purpose and contents of the study and all women signed written consent to participate in the study.

As previously published by Sonmez et al , BT+IVES succeeded to reduce mean incontinence episodes from 4.40±3.43 to 0.70±0.57 after treatment in the active comparator group while mean incontinence episodes was reduced from 4.15±1.67 to 2.68±1.66 after treatment in the control group (BT). Considering a 50% or greater improvement in incontinence episodes in the referred study, the optimum sample size should be 18 cases in each arm with a level of significance of 95% (α=5%), a power of 95% (ß=0.05) . Taking into account possible withdrawals which was assumed to be about 10% of the number of patients, a total of 40 women (20 women for each group) were calculated for this study. Sample size calculation was performed by the physician using G*Power 3.1 Statistical Power Analysis for Microsoft Windows and Mac. Statistics.

To investigators recruited women with complaints of OAB who were referred to the Urogynecological Rehabilitation Unit and other related outpatient clinics. Women over the age of 18 with the clinical diagnosis of idiopathic OAB, and who could able to give written informed consent and understand the procedures were included in this study. The criteria for exclusion were as follows. Women who had stress urinary incontinence; a history of PTNS and/or TTNS for OAB within 6 months; urogynecological surgery within 3 months; current vulvovaginitis or urinary tract infections or malignancy; pregnancy; cardiac pacemaker or implanted defibrillator; anatomic or posttraumatic malformations/skin disorders of tibial nerve region on inner ankle that can not allow to apply the electrodes; the strength of PFM less than 3/5 (graded as modified Oxford scale, min:0-max:5); the pelvic organ prolapse quantification (POP-Q) (stage 2 or more); neurogenic bladder; the peripheral or central neurologic pathology; ultrasonographic evidence of post-void residual urine volume more than 100 ml were excluded.

Women with idiopathic OAB were recruited for eligibility and of them who fulfilled the inclusion/exclusion criteria were included for this study. Antimuscarinic naive women were included in Group 1 (n:20), and women resistant to anti-muscarinic agents were included in Group 2 (n:20). Both groups received BT plus TTNS.

Group 1: Antimuscarinic Naive (AM-N) None of the women had previously taken anti-muscarinic agents and oral ß3 adrenoreceptor agonist (mirabegron) in this group.

Group 1: Antimuscarinic Refractory (AM-R) Women with idiopathic OAB refractory to anti-muscarinic agents and oral ß3 adrenoreceptor agonist (mirabegron) when 2 or more were administered for at least 6 weeks each and failure was due to lack of efficacy with or without side effects were included in this group.

Bladder Training (BT) All women were informed about BT that consisted of four stages and lasted for 30 minutes. Then, it was given as a written brochure to be implemented as a home program. At the first stage, the women were familiarized with the location of the PFM and the pelvic anatomy and pathophysiology. After that information session, squeezing the PFM was shown in practice at least once to use in the urgency suppression strategies via digital palpation technique. The second stage including urgency suppression strategies was aimed to delay urination, inhibit detrusor contraction, and prevent urgency by squeezing the PFM several times on a row, breathing deeply, giving their attention to another job for a while, and self-motivating. In the third stage, a timed voiding program was started. It was carried out in 2 steps: a timed voiding and increasing the time between urination considering the voiding diary. At the last stage, the women were encouraged to continue BT.

Transcutaneous tibial nerve stimulation (TTNS) Two self-adhesive surface electrodes were positioned according to the protocol used by Booth et al and Shreiner et al, with the negative electrode 2 cm behind the medial malleolus and positive electrode 10 cm proximal to it. Correct positioning was determined by noting a hallux reaction (plantar flexion of great toe or fanning of all toes). The stimulation protocol was delivered at fixed of 20 Hz and pulse width of 200 ms in continous mode in accordance with PTNS stimulation protocol. The intensity level of the stimulation current (range 0-50 mA) was determined once correct positioning was established, according to the comfort level of the subject. TTNS sessions were performed two times in a week, for 6 weeks. Every session lasted 30 minutes. The intervention comprised a 12 session treatment program of TTNS.

TTNS sessions were performed by an experienced urogynecological rehabilitation nurse in all groups. During the treatment, all women were advised to continue the medical treatment which was not related to incontinence. Participants were asked to fill in a one-day bladder diary biweekly to continue the timed voiding program, which is part of BT in two groups. Compliance with the BT was achieved with the daily checklist during 6 weeks and the bladder diaries of women were checked biweekly to rearrange the timed voiding program. Women who did not fill more than 20% of the daily checklist and who missed any therapy sessions for two groups were excluded from the study.

Evaluation Parameters The primary outcome measure was accepted as the improvement in incontinence episodes (positive response rate), according to literature . To determine positive response rate, reduction in incontinence episodes was collected from the 3-day bladder diary. Women with ≥a 50% reduction in incontinence episodes were considered positive responders. Furthermore, the severity of incontinence, PFM strength, symptom severity, frequency of voiding, nocturia, number of pads as well as QoL were secondary outcome measures. The 24-hour pad test was carried out to evaluate the severity of incontinence. Overactive Bladder Questionnaire (OAB-V8) was used to evaluate the symptom severity in patients with OAB in this study. The OAB-V8 consists of 8 questions in which the patients can be classified with respect to the symptom severity: none (0), very little (1), a little (2), quite a few (3), very (4), and too many (5). The total score ranges from 0-40. The frequencies of voiding, nocturia, and the number of pads used were collected from the 3-day bladder diary. The Quality of Life-Incontinence Impact Questionnaire (IIQ7) was used to assess specific QoL related to incontinence. In addition, cure-improvement rate and treatment satisfaction were evaluated. In a 24-hour pad test, amount of urine that was under 1.3 gr was considered as a cure. The improvement rate was assessed in terms of 50% and more reduction in wet weight compared to baseline measurements in the 24-hour pad test . Women evaluated the change in their urinary incontinence on a 5-point Likert scale (5, very satisfied; 1, very unsatisfied). All the evaluation tests were performed by another physician who was blinded to the groups in the initial visit and at the end of the treatment (8th week), except for the positive response rate, cure/improvement rate, and the treatment satisfaction parameters which were evaluated only at the 8th week.

Statistics SPSS17.0 software (SPSS, Chicago, IL) was used for the statistical analysis. In each group, measurable parameters were tested with the Kolmogorov-Smirnov test for the evaluation of normal distribution. Because the distributions were not normal, non-parametric tests were used in the statistical evaluation. Mann-Whitney U-test and χ2 test were used for inter-group comparisons. Wilcoxon tests were used for intra-group comparison of parameters at different point of times. P<0.05 was accepted as statistically significant.

ELIGIBILITY:
Inclusion Criteria:

1. Women 18 years and older with clinically idiopathic OAB
2. Having the ability to give written informed consent
3. Ability to understand procedures

Exclusion Criteria:

1. Presence of active vaginal or urinary tract infection or malignancy
2. Pregnancy or intention to become pregnant during the study
3. History of neurogenic bladder, peripheral or central neurological pathology
4. Presence of Grade 2 and higher pelvic organ prolapse (POP) according to the International Continence Society (ICS)
5. Having undergone urogynecological surgery in the last 3 months
6. Women with stress urinary incontinence
7. History of PTNS and/or TTNS for OAB in the past 6 months
8. Presence of a pacemaker or implanted defibrillator
9. Presence of anatomical or post-traumatic malformations / skin disorders of the tibial nerve region of the inner ankle that do not allow the application of electrodes
10. PTK strength less than 3/5 (rated as modified Oxford scale, min: 0-max: 5)
11. Ultrasonographic evidence of a postvoid residual urine volume greater than 100 ml

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 40 (Estimated)
Dates: Start 2023-01-01 (Estimated); Primary Completion 2023-06-01 (Estimated); Study Completion 2023-06-30 (Estimated)

PRIMARY OUTCOMES:
İmprovement in incontinence episodes | 6 months
  To determine positive response rate, reduction in incontinence episodes was collected from the 3-day bladder diary. Women with ≥a 50% reduction in incontinence episodes were considered positive responders

SECONDARY OUTCOMES:
Severity of incontinence | 6 months
  The 24-hour pad test and Overactive Bladder Questionnaire (OAB-V8) was carried out to evaluate the severity of incontinence. The OAB-V8 consists of 8 questions in which the patients can be classified with respect to severity of incontinence: none (0), very little (1), a little (2), quite a few (3), very (4), and too many (5). The total score ranges from 0-40.
The frequencies of voiding | 6 months
  TThe frequencies of voiding, used were collected from the 3-day bladder diary.
Cure-improvement rate | 6 months
  In a 24-hour pad test, amount of urine that was under 1.3 gr was considered as a cure. The improvement rate was assessed in terms of 50% and more reduction in wet weight compared to baseline measurements in the 24-hour pad test.
Change in their urinary incontinence | 6 months
  Women evaluated the change in their urinary incontinence on a 5-point Likert scale (5, very satisfied; 1, very unsatisfied)
Nocturia | 6 months
  Nocturia, used were collected from the 3-day bladder diary.
The number of pads | 6 months
  The number of pads, used were collected from the 3-day bladder diary.
The Quality of Life | 6 months
  The Quality of Life-Incontinence Impact Questionnaire (IIQ7) was used to assess specific QoL related to incontinence. The form consists of 7 questions. In the form, the patients had no complaints (0); less (1); middle (2); many (3); graded as. The total score ranges from 0 to 21. A lower score indicates less quality of life impact.
Treatment satisfaction | 6 months
  A 5-point "treatment satisfaction scale" was used for treatment satisfaction. (1, not at all satisfied 5, very satisfied). A lower score indicates less treatment satisfaction.

CONTACTS AND LOCATIONS:
Locations (1):
- Pamukkale University, Denizli, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Scaldazza CV, Morosetti C, Giampieretti R, Lorenzetti R, Baroni M. Percutaneous tibial nerve stimulation versus electrical stimulation with pelvic floor muscle training for overactive bladder syndrome in women: results of a randomized controlled study. Int Braz J Urol. 2017 Jan-Feb;43(1):121-126. doi: 10.1590/S1677-5538.IBJU.2015.0719. PMID 28124534
- [Background] Kasman A, Stave C, Elliott CS. Combination therapy in overactive bladder-untapped research opportunities: A systematic review of the literature. Neurourol Urodyn. 2019 Nov;38(8):2083-2092. doi: 10.1002/nau.24158. Epub 2019 Sep 4. PMID 31483070
- [Background] Wang S, Lv J, Feng X, Lv T. Efficacy of Electrical Pudendal Nerve Stimulation versus Transvaginal Electrical Stimulation in Treating Female Idiopathic Urgency Urinary Incontinence. J Urol. 2017 Jun;197(6):1496-1501. doi: 10.1016/j.juro.2017.01.065. Epub 2017 Jan 31. PMID 28153510
- [Background] La Rosa VL, Platania A, Ciebiera M, Garzon S, Jedra R, Ponta M, Buttice S. A comparison of sacral neuromodulation vs. transvaginal electrical stimulation for the treatment of refractory overactive bladder: the impact on quality of life, body image, sexual function, and emotional well-being. Prz Menopauzalny. 2019 Jun;18(2):89-93. doi: 10.5114/pm.2019.86834. Epub 2019 Jun 28. PMID 31485205
- [Background] Firinci S, Yildiz N, Alkan H, Aybek Z. Which combination is most effective in women with idiopathic overactive bladder, including bladder training, biofeedback, and electrical stimulation? A prospective randomized controlled trial. Neurourol Urodyn. 2020 Nov;39(8):2498-2508. doi: 10.1002/nau.24522. Epub 2020 Sep 22. PMID 32960999
- [Background] Yildiz N, Alkan H, Sarsan A. Efficacy of intravaginal electrical stimulation added to bladder training in women with idiopathic overactive bladder: A prospective randomized controlled trial. Int Braz J Urol. 2021 Nov-Dec;47(6):1150-1159. doi: 10.1590/S1677-5538.IBJU.2021.0161. PMID 34469668
- [Background] Yildiz N, Alkan H, Findikoglu G. Efficacy of intravaginal electrical stimulation with different treatment frequency in women with refractory idiopathic overactive bladder. Int Braz J Urol. 2022 Jul-Aug;48(4):662-671. doi: 10.1590/S1677-5538.IBJU.2021.0837. PMID 35363455
- [Background] Bo K, Frawley HC, Haylen BT, Abramov Y, Almeida FG, Berghmans B, Bortolini M, Dumoulin C, Gomes M, McClurg D, Meijlink J, Shelly E, Trabuco E, Walker C, Wells A. An International Urogynecological Association (IUGA)/International Continence Society (ICS) joint report on the terminology for the conservative and nonpharmacological management of female pelvic floor dysfunction. Int Urogynecol J. 2017 Feb;28(2):191-213. doi: 10.1007/s00192-016-3123-4. Epub 2016 Dec 5. PMID 27921161
- [Background] Lee HE, Cho SY, Lee S, Kim M, Oh SJ. Short-term Effects of a Systematized Bladder Training Program for Idiopathic Overactive Bladder: A Prospective Study. Int Neurourol J. 2013 Mar;17(1):11-7. doi: 10.5213/inj.2013.17.1.11. Epub 2013 Mar 31. PMID 23610706
- [Background] Berghmans B, van Waalwijk van Doorn E, Nieman F, de Bie R, van den Brandt P, Van Kerrebroeck P. Efficacy of physical therapeutic modalities in women with proven bladder overactivity. Eur Urol. 2002 Jun;41(6):581-7. doi: 10.1016/s0302-2838(02)00178-1. PMID 12074773
- [Background] Wang AC, Wang YY, Chen MC. Single-blind, randomized trial of pelvic floor muscle training, biofeedback-assisted pelvic floor muscle training, and electrical stimulation in the management of overactive bladder. Urology. 2004 Jan;63(1):61-6. doi: 10.1016/j.urology.2003.08.047. PMID 14751349
- [Background] Berghmans LC, Hendriks HJ, De Bie RA, van Waalwijk van Doorn ES, Bo K, van Kerrebroeck PE. Conservative treatment of urge urinary incontinence in women: a systematic review of randomized clinical trials. BJU Int. 2000 Feb;85(3):254-63. doi: 10.1046/j.1464-410x.2000.00434.x. PMID 10671878
- [Background] Abdelbary AM, El-Dessoukey AA, Massoud AM, Moussa AS, Zayed AS, Elsheikh MG, Ghoneima W, Abdella R, Yousef M. Combined Vaginal Pelvic Floor Electrical Stimulation (PFS) and Local Vaginal Estrogen for Treatment of Overactive Bladder (OAB) in Perimenopausal Females. Randomized Controlled Trial (RCT). Urology. 2015 Sep;86(3):482-6. doi: 10.1016/j.urology.2015.06.007. Epub 2015 Jun 30. PMID 26135813
- [Background] Yamanishi T, Yasuda K, Sakakibara R, Hattori T, Suda S. Randomized, double-blind study of electrical stimulation for urinary incontinence due to detrusor overactivity. Urology. 2000 Mar;55(3):353-7. doi: 10.1016/s0090-4295(99)00476-8. PMID 10699609
- [Background] O'Sullivan R, Karantanis E, Stevermuer TL, Allen W, Moore KH. Definition of mild, moderate and severe incontinence on the 24-hour pad test. BJOG. 2004 Aug;111(8):859-62. doi: 10.1111/j.1471-0528.2004.00211.x. PMID 15270937
- [Background] Tarcan T, Mangır N, Özgür MÖ, Akbal C. OAB-V8 Overactive Bladder Questionnaire Validation Study. (Turkish) Üroloji Bülteni 2012;21:113-116. http://www.kontinansdernegi.org/userfiles/media/kontinans.galenos.com.tr/oab-v8-asiri-aktif-mesane-sorgulama-formu.pdf
- [Background] Acquadro C, Kopp Z, Coyne KS, Corcos J, Tubaro A, Choo MS, Oh SJ. Translating overactive bladder questionnaires in 14 languages. Urology. 2006 Mar;67(3):536-40. doi: 10.1016/j.urology.2005.09.035. PMID 16527574
- [Background] Cam C, Sakalli M, Ay P, Cam M, Karateke A. Validation of the short forms of the incontinence impact questionnaire (IIQ-7) and the urogenital distress inventory (UDI-6) in a Turkish population. Neurourol Urodyn. 2007;26(1):129-33. doi: 10.1002/nau.20292. PMID 17083117
- [Background] Barroso JC, Ramos JG, Martins-Costa S, Sanches PR, Muller AF. Transvaginal electrical stimulation in the treatment of urinary incontinence. BJU Int. 2004 Feb;93(3):319-23. doi: 10.1111/j.1464-410x.2004.04608.x. PMID 14764129
- [Background] Amaro JL, Gameiro MO, Kawano PR, Padovani CR. Intravaginal electrical stimulation: a randomized, double-blind study on the treatment of mixed urinary incontinence. Acta Obstet Gynecol Scand. 2006;85(5):619-22. doi: 10.1080/00016340500495058. PMID 16752244
- [Background] Wang AC, Chih SY, Chen MC. Comparison of electric stimulation and oxybutynin chloride in management of overactive bladder with special reference to urinary urgency: a randomized placebo-controlled trial. Urology. 2006 Nov;68(5):999-1004. doi: 10.1016/j.urology.2006.05.038. PMID 17113893
- [Background] Sonmez R, Yildiz N, Alkan H. Efficacy of percutaneous and transcutaneous tibial nerve stimulation in women with idiopathic overactive bladder: A prospective randomised controlled trial. Ann Phys Rehabil Med. 2022 Jan;65(1):101486. doi: 10.1016/j.rehab.2021.101486. Epub 2021 Nov 11. PMID 33429090
- [Background] Burkhard FC, Bosch JLHR, Cruz F, Lemack GE, Nambiar AK, Thiruchelvam N, et al. The European Association of Urology (EAU) Guidelines. EAU Guidelines on urinary incontinence in adults. In: EAU Guidelines, 2018 (Internet). Available online at: http://uroweb.org/guideline/urinary-incontinence/
- [Background] Gormley EA, Lightner DJ, Faraday M, Vasavada SP; American Urological Association; Society of Urodynamics, Female Pelvic Medicine. Diagnosis and treatment of overactive bladder (non-neurogenic) in adults: AUA/SUFU guideline amendment. J Urol. 2015 May;193(5):1572-80. doi: 10.1016/j.juro.2015.01.087. Epub 2015 Jan 23. PMID 25623739
- [Background] Booth J, Hagen S, McClurg D, Norton C, MacInnes C, Collins B, Donaldson C, Tolson D. A feasibility study of transcutaneous posterior tibial nerve stimulation for bladder and bowel dysfunction in elderly adults in residential care. J Am Med Dir Assoc. 2013 Apr;14(4):270-4. doi: 10.1016/j.jamda.2012.10.021. Epub 2012 Nov 30. PMID 23206722
- [Background] Manriquez V, Guzman R, Naser M, Aguilera A, Narvaez S, Castro A, Swift S, Digesu GA. Transcutaneous posterior tibial nerve stimulation versus extended release oxybutynin in overactive bladder patients. A prospective randomized trial. Eur J Obstet Gynecol Reprod Biol. 2016 Jan;196:6-10. doi: 10.1016/j.ejogrb.2015.09.020. Epub 2015 Oct 20. PMID 26645117
- [Background] Schreiner L, dos Santos TG, Knorst MR, da Silva Filho IG. Randomized trial of transcutaneous tibial nerve stimulation to treat urge urinary incontinence in older women. Int Urogynecol J. 2010 Sep;21(9):1065-70. doi: 10.1007/s00192-010-1165-6. Epub 2010 May 11. PMID 20458465
- [Background] Ramirez-Garcia I, Blanco-Ratto L, Kauffmann S, Carralero-Martinez A, Sanchez E. Efficacy of transcutaneous stimulation of the posterior tibial nerve compared to percutaneous stimulation in idiopathic overactive bladder syndrome: Randomized control trial. Neurourol Urodyn. 2019 Jan;38(1):261-268. doi: 10.1002/nau.23843. Epub 2018 Oct 12. PMID 30311692